CLINICAL TRIAL: NCT04462484
Title: Study Protocol of a Randomized Controlled Trial of an Online Self-Care Training Programme to Reduce Burnout and Promote Work Engagement in Clinical Psychologists: MAGO Study
Brief Title: Online Self-care Training Program (MAGO Study)
Acronym: MAGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: University of Chile (Other)
Responsible Party: Principal Investigator, Sabrina Cipolletta, Associate Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-12/2020
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Occupational Burnout
Keywords: burnout; self-care; online program; telepsychology
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: MAGO is a parallel, two-armed randomized controlled trial with three assessment points (baseline, post-intervention, and six-month follow-up). Participants will be randomized for the program or a no-treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention
- Intervention group (Experimental): Videoconference
  Interventions: Behavioral: videoconference

INTERVENTIONS:
Behavioral: videoconference — The intervention is a person-directed, individual, primary occupational intervention. It will be carried out via videoconference in six sessions of 45 minutes (on a weekly basis). Through guided dialogue, individual difficulties and opportunities of each subject will be examined in order to gain self-awareness of personal characteristics (strengths, limitations, maximum workload capacity) in their particular set of job demands and resources. Participants are encouraged to adopt the set of self-care strategies in each dimension, adapting them to their specific context. Activities will be carried out in Spanish by the researcher.
  Arms: Intervention group

SUMMARY:
This study aims to determine the efficacy of MAGO (Online Self-care Training Program for Psychologists), a person-directed, individual, occupational intervention via videoconference in six sessions on a weekly basis. By promoting self-care behaviors, it is expected to reduce burnout levels and to increase work engagement in clinical psychologists working in Chile.

DETAILED DESCRIPTION:
Clinical psychologists are susceptible to develop burnout as a result of facing consistently emotionally taxing job demands and a high requirement for empathy. Implementing self-care behaviors can help to prevent negative consequences of work stress and the promotion of positive outcomes such as optimal professional functioning and enhanced well-being in psychologists.

The intervention is a person-directed, individual, primary occupational intervention. It will be carried out via videoconference in six weekly sessions of 45 minutes. MAGO is a program derived from Self-care Assessment for Psychology (SCAP). From a preventive perspective on self-care, items represent strategies or behaviors that may be integrated into one's professional and personal life on a more ongoing and proactive basis to promote well-functioning.

Chile has presented a slow but progressive development of e-mental health research, and Internet-based interventions are at an early stage of development in this country. Using videoconference and web-delivered questionnaires are crucial in reaching psychologists considering problems such as long distances of transportation and a tiny budget for mental health. Nevertheless, Chile scores 52 in the Global Connectivity Index, while digital technologies are highly utilized across all social strata.

ELIGIBILITY:
Inclusion Criteria:

* Chilean psychologists
* Currently working in the public sector in Chile
* Available to attend to six online sessions
* Willing to voluntarily participate

Exclusion Criteria:

* Subjects participating in psychotherapy as clients
* High scores for depression or anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-02-13 (Actual); Study Completion 2022-02-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline occupational burnout | 8 weeks and 6 months.
  Maslach Burnout Inventory for human services (MBI-HSS) is comprised of 22 items to evaluate emotional exhaustion (EE), depersonalization (DP), and personal fulfillment (PF). Total score ranges from 0 to 132, with higher scores indicating more occupational burnout.
Change from baseline work engagement | 8 weeks and 6 months.
  Utrecht Work Engagement (UWES-17) is comprised of 17 items. Total score ranges from 0 to 102, with higher scores indicating more work engagement.

SECONDARY OUTCOMES:
Change from baseline self-care behaviors | 8 weeks and 6 months.
  Self-Care Assessment for Psychologists (SCAP) is comprised of 21 items. Total score ranges from 21 to 147, with higher scores indicating higher frequency of self-care behaviors.
Change from baseline general health | 8 weeks and 6 months.
  General Health Questionnaire (GHQ-12) is comprised of 12 items. Total score ranges from 0 to 12, with higher scores indicating lower levels general health.
Change from baseline perceived social support | Baseline, 8 weeks, 6 months.
  Multidimensional Scale of Perceived Social Support (MSPSS) is comprised of 12 items. Total score ranges from 12 to 84, with higher scores indicating higher levels of perceived social support.
Change from baseline depression symptoms | 8 weeks and 6 months.
  Beck Depression Inventory (BDI-II) is comprised of 21 items. Total score ranges from 0 to 63, with higher scores indicating higher levels of depressive symptomatology.
Change from baseline anxiety symptoms | 8 weeks and 6 months.
  Beck Anxiety Inventory (BAI) is comprised of 21 items. Total score ranges from 0 to 63 with higher scores indicating higher levels of anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Cipolletta, PhD, Study Director — University of Padova; Caterina Novara, PhD, Study Director — University of Padova
Locations (1):
- Universidad de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dorociak KE, Rupert PA, Bryant FB, Zahniser E. Development of the Professional Self-Care Scale. J Couns Psychol. 2017 Apr;64(3):325-334. doi: 10.1037/cou0000206. Epub 2017 Mar 9. PMID 28277686
- See also: Huawei Global Connectivity Index. (2019) — https://www.huawei.com/minisite/gci/assets/files/gci_2019_whitepaper_en.pdf?v=20191217v2

DOCUMENTS (1):
  • Informed Consent Form (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT04462484/ICF_001.pdf